CLINICAL TRIAL: NCT01072253
Title: Quality of Life of Eye Amputated Patients in Denmark
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Velux Fonden (Other); The Danish Eye Research foundation (Unknown)
Other Study IDs: Velux270479
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Eye Cancer; Painful Blind Eye; Panophthalmia; Traumas
MeSH Terms: conditions — Eye Neoplasms; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- eye amputated: lost an eye
  Interventions: Procedure: eye amputation

INTERVENTIONS:
Procedure: eye amputation

SUMMARY:
The purpose of this study is to evaluate eye amputated patients health related quality of life, perceived stress, self-rated health, labour marked participation and socio-economic position.

The investigators hypothesis is that quality of life, perceived stress and self- rated health of many eye amputated patients are drastically changed. Eye amputation has a marked negative influence on labour marked participation and socio-economic position of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were operation for evisceration, enucleation, orbital exenteration or secondary implantation of an orbital implant during the period 1996-2003. 267 patients were in 2005 invited to a clinical investigation and of those 173 accepted.
* Included in this study were patients who came to the clinical investigation, who accepted to receive questionnaires and were alive in 2008.

Exclusion Criteria:

* Dead
* Below 18 years
* Left the country
* Living at Greenland or the Faeroe Islands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: eye clinic Rigshospitalet, Denmark. Rigshospitalet is a public, regionalized and national specialized hospital with a recruitment area of Eastern Denmark (approximately 2 million people). Nearly all cases of eye amputation and cancer in the eye region in Eastern Denmark are performed at Rigshospitalet
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Marie Louise R Rasmussen, MD, Principal Investigator — University of Copenhagen; Peter B Toft, MD, DMSc, Study Director — University of Copenhagen
Locations (1):
- Department of Neuroscience and pharmacology, section of eye pathology, Copenhagen, Seland, Denmark

REFERENCES:
- [Background] Roed Rasmussen ML, Prause JU, Johnson M, Toft PB. Phantom eye syndrome: types of visual hallucinations and related phenomena. Ophthalmic Plast Reconstr Surg. 2009 Sep-Oct;25(5):390-3. doi: 10.1097/IOP.0b013e3181b54b06. PMID 19966655
- [Background] Rasmussen ML, Prause JU, Johnson M, Kamper-Jorgensen F, Toft PB. Review of 345 eye amputations carried out in the period 1996-2003, at Rigshospitalet, Denmark. Acta Ophthalmol. 2010 Mar;88(2):218-21. doi: 10.1111/j.1755-3768.2008.01435.x. Epub 2008 Dec 24. PMID 19141150